CLINICAL TRIAL: NCT01348035
Title: Efficacy Study of Long-term Water Intake on the Progression of Autosomal Dominant Polycystic Kidney Disease (ADPKD).
Brief Title: Efficacy Study of Water Drinking on PKD Progression.
Acronym: ESWP
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Eiji Higashihara, MD, Professor, Kyorin University
Other Study IDs: KYR-003-PKD
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease; Disease Progression
Keywords: Autosomal Dominant Polycystic Kidney Disease.; Arginine vasopressin; Total Kidney Volume; Glomerular Filtration Rate
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Disease Progression; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Water Load Group: Water load group: 2.5 ~ 3 L water intake daily for 12 months (50ml/Kg body weight/day). When large amount water intake is not sustainable, patients can reduce the amount of water intake to the levels as much as large he or she can sustain.
- Non-Water Loaded Group: Non-water load group: The patients are free to access water intake, as they like.

SUMMARY:
This is a prospective 5-year study to compare the change in total kidney volume (TKV) before and after tolvaptan therapy, as the primary endpoint, in patients with ADPKD.

DETAILED DESCRIPTION:
Tolvaptan was approved in Japan for the treatment of autosomal dominant polycystic kidney disease (ADPKD) in March 2014. This is a prospective 5-year study to compare the change in total kidney volume (TKV) before and after tolvaptan therapy, as the primary endpoint, in patients with ADPKD. Study results will be summarized, analyzed, and compiled into a research paper at 3 years (data cut-off, March 31, 2018) and at 5 years (data cut-off, March 31, 2020)

ELIGIBILITY:
Inclusion Criteria:

* The patients with ADPKD
* The patients who consent to the study protocol
* Estimated glomerular filtration rate (eGFR) or Creatinine Clearance greater than 50ml/min/1.73m2

Exclusion Criteria:

* Patients who might be danger to drink large amount of water such as having heart failure or past history of cerebrovascular or cardiovascular disorders.
* The patients who take habitual medication which affects the AVP action such as selective serotonin reuptake inhibitors (SSRI ), tricyclic antidepressants or diuretics.
* The patients who is considered inappropriate by physicians.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who visit Kyorin University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Total kidney volume (TKV) measured by magnetic resonance imaging (MRI). | One year (12 months) and pre-study period.
  The relationship between urine volume (and urine osmolality) and change of TKV. TKV slopes are compared between pre-study and study period.

SECONDARY OUTCOMES:
Glomerular filtration rate (GFR) estimated by plasma creatinine and cystatin C. | One year (12 months)
  The relationship between urine volume (and urine osmolality) and change of GFR.
Plasma arginine vasopressin (AVP, Copeptin) level. | 4-8-12 months
  The relationship between urine volume (osmolality) and plasma AVP.
Quality of life (QOL) questionnaire. | 4-8-12 months
  The relationship between QOL and urine volume.

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Higashihara, M.D., Principal Investigator — Kyorin University
Locations (1):
- Department of Urology, Kyorin University Hospital, Mitaka, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No